CLINICAL TRIAL: NCT06998901
Title: Effect of FIFA 11+ Kids Training Programme on Injury Prevention and Athletic Performance in U-14 Basketball Players
Brief Title: The Effect of FIFA 11+ Kids Training Programme on Injury Prevention and Athletic Performance in U-14 Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monira Aldhahi (Other)
Responsible Party: Sponsor-Investigator, Monira Aldhahi, Associate Professor, Princess Nourah Bint Abdulrahman University
Organization: Princess Nourah Bint Abdulrahman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PNU1
Record Dates: First submitted 2025-05-21; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ Kids Training Intervention Group (Experimental): Participants in this arm will receive the FIFA 11+ Kids training program in addition to their regular basketball practice. The program consists of structured neuromuscular warm-up exercises designed to improve balance, coordination, strength, and overall movement control. It will be implemented over a period of 7 weeks, with sessions conducted four times per week, each lasting approximately 15-20 minutes. The exercises are age-appropriate and follow a progressive format to enhance athletic performance and reduce injury risk in youth athletes.
  Interventions: Other: FIFA 11+ Kids training program
- Standard Basketball Training Control Group (No Intervention): Participants in this arm will continue with their regular basketball training routine without the addition of the FIFA 11+ Kids program. The training will follow the standard practice schedule implemented by their coaches, focusing on technical skills, game strategy, and general physical conditioning. No structured neuromuscular warm-up or injury-prevention program will be introduced during the intervention period. This arm will serve as a comparison to evaluate the effects of the FIFA 11+ Kids training program on athletic performance and movement quality.

INTERVENTIONS:
Other: FIFA 11+ Kids training program — Participants in this arm will receive the FIFA 11+ Kids training program in addition to their regular basketball practice. The program consists of structured neuromuscular warm-up exercises designed to improve balance, coordination, strength, and overall movement control. It will be implemented over a period of 7 weeks, with sessions conducted four times per week, each lasting approximately 15-20 minutes. The exercises are age-appropriate and follow a progressive format to enhance athletic performance and reduce injury risk in youth athletes.
  Arms: FIFA 11+ Kids Training Intervention Group

SUMMARY:
This study aims to evaluate the effects of the FIFA 11+ Kids training program on the athletic performance and Functional Movement Screen (FMS) scores of under-14 male basketball players. A total of 40 participants will be randomly assigned to either a training group or a control group. The training group will follow the FIFA 11+ Kids program for seven weeks, while the control group will continue with regular basketball training. Performance tests-including vertical jump, sprint, agility, standing long jump, and FMS-will be used to assess the impact of the intervention. The goal is to determine whether the FIFA 11+ Kids program can enhance athletic performance and movement quality in youth basketball players.

DETAILED DESCRIPTION:
This study is designed to assess the impact of the FIFA 11+ Kids training program on key athletic performance indicators and movement quality in under-14 male basketball players. The research will involve a randomized controlled trial in which participants will be divided into two groups: an intervention group that undergoes the FIFA 11+ Kids program in addition to their regular basketball training, and a control group that continues with standard basketball training only.

The intervention will be implemented over a period of seven weeks, with sessions held four times per week, each lasting approximately 15 to 20 minutes. The program focuses on improving neuromuscular control, balance, and strength through age-appropriate exercises.

Pre- and post-intervention assessments will include standardized athletic performance tests (vertical jump, sprint, agility, and standing long jump) and movement quality evaluation using the Functional Movement Screen (FMS). The study aims to determine whether short-term implementation of the FIFA 11+ Kids program can produce measurable improvements, particularly in explosive power and movement efficiency. Results will guide recommendations for integrating injury-prevention programs into youth basketball training.

ELIGIBILITY:
Inclusion Criteria:

* Male basketball players aged 11 to 13 years
* Actively participating in organized basketball training at least 3 times per week
* No prior exposure to the FIFA 11+ Kids training program
* Able to provide informed consent from a parent or legal guardian
* Physically able to perform the required exercises and tests included in the study

Exclusion Criteria:

* Current musculoskeletal injury or medical condition that limits participation in physical activity
* History of surgery or major injury in the past 6 months
* Diagnosis of any neurological, cardiovascular, or respiratory disorder affecting performance
* Participation in another structured injury prevention or neuromuscular training program during the study period
* Inability to understand or follow instructions for the training or testing procedures

Ages: 7 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen Test Protocol | From enrollment to the end of treatment at 7 weeks
  The Functional Movement Screen (FMS) is used to assess fundamental movement patterns, mobility, and stability. It consists of seven test components: deep squat, hurdle step, inline lunge, shoulder mobility, active straight leg raise, trunk stability push-up, and rotary stability. Each movement is scored on a scale from 0 to 3, with a maximum possible total score of 21. The test is administered by trained personnel following standardized procedures, and the total FMS score is used to evaluate overall movement quality and identify potential risk for injury.
Pro-Agility Test (5-10-5 Shuttle Run): | From enrollment to the end of treatment at 7 weeks
  Agility is measured using a shuttle run between markers set 4.57 meters apart. Participants complete two timed trials, and the fastest time is used for analysis.
Countermovement Jump Test: | From enrollment to the end of treatment at 7 weeks
  Vertical jump performance is assessed using a waist-worn accelerometer. Participants perform two maximal vertical jumps, and the highest value is recorded for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy and Rehabilitation, Faculty of Medicine, Tekirdağ Namık Kemal University, Tekirdağ, Turkey,, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided